CLINICAL TRIAL: NCT00587925
Title: A Pilot Study of Bone Mineral Density in Postmenopausal Women After Treatment for Breast Cancer
Brief Title: Study of Bone Mineral Density in Postmenopausal Women After Treatment for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Gabriella D'Andrea, MD, Memorial Sloan-Kettering Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-024
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Bone Density

ARMS (1):
- 1 (Experimental): Bone Mineral Density
  Interventions: Other: Bone Mineral Density

INTERVENTIONS:
Other: Bone Mineral Density — Clinic visits twice during the first 2 years of the study with medical care directed by your treating doctor.BMD is measured by an X-ray test. The most common type of BMD testing is by energy x-ray absorptiometry (DEXA). Usually BMD is measured every other year, but to closely monitor women on this study, the BMD will be evaluated more often. The BMD will be measured 3 times (baseline, 12 months and 24 months) on this study. Study blood work is obtained three times (baseline, 6 months, and 12 months). Blood (about 3 teaspoons).

SUMMARY:
Bone Mineral Density (BMD) as measured by X-ray shows the amount of calcium in the bone. Low BMD may reflect osteoporosis, a condition where there is an increased risk of fracture. Women who have gone through menopause have a higher risk of getting osteoporosis because they lose calcium from their bones much faster than younger women. Women with breast cancer may have an additional risk for getting osteoporosis because of the effects of their treatment with chemotherapy. The purpose of this study is to see what levels of BMD post-menopausal women with breast cancer have, and to see if the level of BMD changes during a women's treatment after her surgery. This trial studies changes in BMD and markers of bone activity in women receiving treatment for early stage breast cancer.

DETAILED DESCRIPTION:
Breast cancer patients may be at increased risk for osteoporosis secondary to cancer treatment. The hypothesis of this study is that adjuvant chemotherapy increases the risk of osteoporosis in postmenopausal women. The objective of this pilot study is to describe the effects of chemotherapy on bone mineral density and serum markers of bone metabolism.

There is limited data on the change in bone mineral density due to chemotherapy in postmenopausal women. This prospective study will gather data on the effects of systemic breast cancer therapy on bone mineral density in postmenopausal women receiving adjuvant care for early stage (0, I, II or III) breast cancer. Postmenopausal women are the focus of this study because: (1) they are the largest subgroup of women with breast cancer (2) they are expected to have a rate of BMD loss unless disturbed by disease or medications, unlike the pre and perimenopausal women whose BMD is dramatically affected by changes in hormonal status (3) this group of patients is at greatest risk for acute osteoporotic fractures.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically or cytologically proven diagnosis of breast cancer
* Non-metastatic breast cancer tumor with the diagnosis of Tis, T1-T4, N0-3, M0 (Stage 0, I, II or III breast cancer) by the American Joint Committee on Cancer revised tumor-nodal-metastases staging system (Singletary, JCO 2002). DCIS is allowed, but LCIS (only) is not. Adjuvant care is administered as clinically indicated. Adjuvant treatment decisions are not stipulated in this trial.
* Postmenopausal as defined by last menstrual cycle occurring more than 5 years previously. Women who have had a hysterectomy without bilateral oophorectomy will be considered postmenopausal if greater than 55 years of age. Women who have had a bilateral oophorectomy more than 5 years previously will be considered postmenopausal.
* Chemotherapy Arm: Patients about to begin adjuvant, or neoadjuvant, treatment with Doxorubicin (60mg/m2), Cyclophosphamide (600mg/m2) followed by Paclitaxel (175mg/m2) (AC-T) or Doxorubicin (60mg/m2) for 4 cycles followed by Paclitaxel (175mg/m2) for 4 cycles followed by Cyclophosphamide (600mg/m2) for 4 cycles (A-T-C) administered in the dose dense regimen every 2 weeks with growth
* factor support. The patient may enter this trial within 3 months of initiating adjuvant chemotherapy.
* Observation Arm: Patients begin adjuvant follow up with expectant monitoring (no systemic therapy). The patient may enter this trial within 2 months of initiating adjuvant care.
* Signed informed consent
* Assessment of the complete blood count and complete biochemical profile must indicate absolute neutrophil count >1000/ul, hemoglobin > 9 g/dl and platelets >100,000/ul and the bilirubin, liver transaminases (AST/ALT) and serum creatinine must be within 2.5 times the institutional upper level of normal at the time of enrollment into the study.

Exclusion Criteria:

* Any metabolic bone disease (including Paget's disease of the bone) other than postmenopausal osteoporosis or osteopenia.
* Use of systemic gonadal hormonal medications or supplements within the past 24 months. Topical vaginal estrogens such as "Estring" or other vaginal estrogenic compounds not associated with systemic absorption are allowed.
* Prior use of tamoxifen or raloxifene is permitted if the medication was discontinued more then 24 months prior to the diagnosis of breast cancer. No adjuvant antiestrogen, antineoplastic, therapies are permitted on study.
* Chronic use of systemic steroids (equivalent of prednisone 5mg daily for more then 3 months) for disease process other than breast cancer chemotherapy premedications or antiemetics. Inhaled steroids are allowed, as is the occasional use of low to moderate dose short pulse steroids.
* History of rheumatoid arthritis, ankylosing spondylitis, hyperparathyroidism, renal osteodystrophy, moderate to severe inflammatory or autoimmune diseases or newly diagnosed thyroid condition requiring titration of medications (stable dose and minor dose modifications of thyroid medications are acceptable). Other exclusionary comorbid conditions include thalassemia, moderate to severe malabsorptive syndromes and HIV. Patients diagnosed with the above conditions or similar comorbid and/or inflammatory diseases associated with changes in BMD either from the disease process or the therapy of such condition(s) during the course of the study will be removed from the study at the point of diagnosis.
* Lobular carcinoma in situ (LCIS) or Stage IV breast cancer and patients with a concurrently active second malignancy other then adequately treated non-melanoma skin cancers or in situ cervical cancer. Patients with non-mammary malignancies, or prior breast cancer, must have been disease free for at least 5 years.
* Participation in other clinical trials that are measuring BMD as a study parameter
* Patients with conditions that are expected to distort BMD reading and make DEXA results unreliable such as bilateral prosthetic hips, extensive degenerative joint disease, or severe calcification of the aorta.
* Patients with concurrent medical or psychiatric conditions, which at the judgment of the consenting investigator, would prevent them from understanding and complying with this clinical trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
To estimate the rate of change in bone mineral density in postmenopausal women undergoing adjuvant chemotherapy with dose dense doxorubicin, cyclophosphamide and paclitaxel (AC-T or A-T-C) for early stage breast cancer. | conclusion of study

SECONDARY OUTCOMES:
To estimate the rate of change in markers of bone metabolism in postmenopausal women undergoing adjuvant chemotherapy with doxorubicin, cyclophosphamide and paclitaxel (AC-T or A-T-C) for early stage breast cancer. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Dandrea, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org